CLINICAL TRIAL: NCT00098748
Title: A Multicenter, Randomized, Double-Blind Placebo-Controlled Trial of a Novel CCR5 Antagonist, UK-427,857, in Combination With Optimized Background Therapy Versus Optimized Background Therapy Alone for the Treatment of Antiretroviral-Experienced, Non CCR5-Tropic HIV-1 Infected Subjects
Brief Title: Trial of Maraviroc (UK-427,857) in Combination With Optimized Background Therapy Versus Optimized Background Therapy Alone for the Treatment of Antiretroviral-Experienced NonCCR5-Tropic HIV-1 Infected Subjects
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4001029
Record Dates: First submitted 2004-12-07; First posted 2004-12-08 (Estimated); Results first posted 2010-10-21 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2010-11

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Maraviroc

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Optimized Background Therapy (OBT); Drug: maraviroc (UK-427,857)
- 2 (Experimental)
  Interventions: Drug: Optimized Background Therapy (OBT); Drug: maraviroc (UK-427,857)
- 3 (Experimental)
  Interventions: Drug: Optimized Background Therapy (OBT)

INTERVENTIONS:
Drug: Optimized Background Therapy (OBT) — OBT (3-6 drugs based on treatment history and resistance testing)
  Arms: 1
Drug: maraviroc (UK-427,857) — maraviroc (UK-427,857) 150 mg taken once daily
  Other Names: Selzentry, Celsentri
  Arms: 1
Drug: Optimized Background Therapy (OBT) — OBT (3-6 drugs based on treatment history and resistance testing)
  Arms: 2
Drug: maraviroc (UK-427,857) — maraviroc (UK-427,857) 150 mg taken twice daily
  Other Names: Selzentry, Celsentri
  Arms: 2
Drug: Optimized Background Therapy (OBT) — OBT (3-6 drugs based on treatment history and resistance testing)
  Arms: 3

SUMMARY:
Maraviroc (UK-427,857), a selective and reversible CCR5 co-receptor antagonist, has been shown to be active in vitro against a wide range of clinical isolates (including those resistant to existing classes). In HIV-1 infected patients in the United States, maraviroc (UK-427,857) is approved for use as part of combination antiretroviral treatment in treatment-experienced and treatment-naive adult subjects. At least 50% of treatment-experienced patients are infected with R5-tropic HIV-1 exclusively. However, even in patients infected with a dual tropic (R5 + X4) phenotype, a large proportion of the virus population still uses CCR5 exclusively. Thus, the purpose of this study is to evaluate the antiretroviral activity, and safety, of maraviroc (UK-427,857) (in combination with other agents) in HIV infected, treatment experienced patients who are failing their current antiretroviral regimen and not infected with R5-tropic virus exclusively. This study will involve more than 200 centers globally to achieve a total randomized subject population of 192 subjects. Patients will be randomly (1:1:1) assigned to one of three groups: Optimized Background Therapy [OBT (3-6 drugs based on treatment history and resistance testing)] + maraviroc (UK-427,857) 150 mg taken once daily, OBT + maraviroc (UK-427,857) 150 mg taken twice daily, or OBT alone. Randomization was stratified by Enfuvirtide use in OBT (yes/no) and Screening HIV-1 RNA level (viral load) (<100,000/≥ 100, 000 copies per milliliter [copies per mL]). The study will enroll over approximately a 9 month period with 48 weeks of treatment. Physical examinations will be performed at study entry, weeks 4, 8, 12, 16, 20, 24, 32, 40 and 48. Blood samples will also be taken at study entry, weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, and 48. Additionally, blood samples will be drawn twice, at least 30 minutes apart, at weeks 2 and 24 for maraviroc (UK-427,857) pharmacokinetic analysis. As part of this clinical study a blood sample will also be taken for non-anonymized pharmacogenetic analysis. Patients will undergo a 12-lead electrocardiogram at study entry, weeks 24 and 48.

DETAILED DESCRIPTION:
(i) Subjects remained on their assigned therapy for 48 weeks, unless the subject was discontinued early for protocol-defined treatment failure or other reasons such as adverse event, loss to follow-up, withdrawal of consent, or death.

(ii) If a subject met the criteria for treatment failure or discontinued for another reason (eg, pregnancy, adverse event) and required an alternative regimen, the subject was followed until the Week 48 visit according to protocol guidelines. The new regimen, selected by the Investigator based on the results of resistance testing at the time of failure, had to be recorded in the CRF.

(iii) Open-label maraviroc (UK-427,857) was provided by the sponsor, until it was commercially available, to subjects who completed 48 weeks of therapy and for whom it was medically appropriate to continue therapy with maraviroc (UK-427,857).

ELIGIBILITY:
Inclusion Criteria:

* Men or women at least 16 years of age (or minimum age as determined by local regulatory authorities)
* HIV-1 RNA viral load of greater than or equal to 5,000 copies/mL
* Stable pre-study antiretroviral regimen, or on no antiretroviral agents, for at least 4 weeks
* Documented genotypic or phenotypic resistance to two of the four antiretroviral drug classes, OR, Antiretroviral-class experience greater than or equal to 3 months (sequential or cumulative) with at least three of the following: One nucleoside or nucleotide reverse transcriptase inhibitor (excluding low-dose ritonavir) and/or enfuvirtide
* Be willing to remain on randomized treatment without any changes or additions to the OBT regimen, except for toxicity management or upon meeting criteria for treatment failure
* A negative urine pregnancy test at the baseline visit for Women of Child Bearing Potential (WOCBP)
* Effective barrier contraception for WOCBP and males

Exclusion Criteria:

* Patients requiring treatment with more than 6 antiretroviral agents (excluding low-dose ritonavir)
* Prior treatment with maraviroc (UK-427,857) or another experimental HIV entry inhibitor for more than 14 days
* Suspected or documented active, untreated HIV-1 related opportunistic infection (OI) or other condition requiring acute therapy
* Treatment for an active opportunistic infection, or unexplained temperature >38.5 degrees Celsius for 7 consecutive days
* Active alcohol or substance abuse sufficient, in the Investigator's judgment, to prevent adherence to study medication and/or follow up
* Lactating women, or planned pregnancy during the trial period
* Significant renal insufficiency
* Previous therapy with a potentially myelosuppressive, neurotoxic, hepatotoxic and/or cytotoxic agent within 30 days prior to randomization or the expected need for such therapy during the study period
* Documented or suspected acute hepatitis or pancreatitis within 30 days prior to randomization
* Significantly elevated liver enzymes or cirrhosis
* Significant neutropenia, anemia or thrombocytopenia
* Malabsorption or an inability to tolerate oral medications
* Symptomatic postural hypotension or severe cardiovascular or cerebrovascular disease
* Certain medications
* Malignancy requiring parenteral chemotherapy that must be continued for the duration of the trial
* R5 virus phenotype only
* No option to use at least one non-nucleoside reverse transcriptase inhibitor or protease inhibitor, or enfuvirtide, based on resistance testing
* Any other clinical condition that, in the Investigator's judgment, would potentially compromise study compliance or the ability to evaluate safety/efficacy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2004-11; Primary Completion 2005-12 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (57):
- United States (34):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Beverly Hills, California
  - Pfizer Investigational Site, Fountain Valley, California
  - Pfizer Investigational Site, Hayward, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Newport Beach, California
  - Pfizer Investigational Site, Oakland, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Union City, California
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, North Miami Beach, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Sarasota, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Vero Beach, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Springfield, Massachusetts
  - Pfizer Investigational Site, Santa Fe, New Mexico
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Brooklyn, New York
  - Pfizer Investigational Site, Manhasset, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Stony Brook, New York
  - Pfizer Investigational Site, The Bronx, New York
  - Pfizer Investigational Site, Huntersville, North Carolina
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Columbia, South Carolina
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Annandale, Virginia
  - Pfizer Investigational Site, Puyallup, Washington
  - Pfizer Investigational Site, Tacoma, Washington
  - Pfizer Investigational Site, Vancouver, Washington
- Australia (5):
  - Pfizer Investigational Site, Darlinghurst, New South Wales
  - Pfizer Investigational Site, Surry Hills, New South Wales
  - Pfizer Investigational Site, Herston, Queensland
  - Pfizer Investigational Site, Carlton, Victoria
  - Pfizer Investigational Site, Melbourne, Victoria
- Belgium (2):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Liège
- Canada (3):
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
- Germany (3):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Cologne
  - Pfizer Investigational Site, Hamburg
- Pfizer Investigational Site, Utrecht, Netherlands
- Spain (5):
  - Pfizer Investigational Site, Elche, Alicante
  - Pfizer Investigational Site, Badalona, Barcelona
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Córdoba, Cordoba
  - Pfizer Investigational Site, Madrid, Madrid
- Pfizer Investigational Site, Zurich, Switzerland
- United Kingdom (3):
  - Pfizer Investigational Site, Brighton
  - Pfizer Investigational Site, Edinburgh
  - Pfizer Investigational Site, London

REFERENCES:
- [Derived] Saag M, Goodrich J, Fatkenheuer G, Clotet B, Clumeck N, Sullivan J, Westby M, van der Ryst E, Mayer H; A4001029 Study Group. A double-blind, placebo-controlled trial of maraviroc in treatment-experienced patients infected with non-R5 HIV-1. J Infect Dis. 2009 Jun 1;199(11):1638-47. doi: 10.1086/598965. PMID 19432546
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4001029&StudyName=Trial%20of%20Maraviroc%20%28UK-427%2C857%29%20in%20Combination%20with%20Optimized%20Background%20Therapy%20Versus%20Optimized%20Background%20Therapy%20Alone%20for%20the%20Tre

RESULTS

PARTICIPANT FLOW:
Groups:
- Maraviroc QD: Maraviroc 150 mg by mouth (PO) once daily (QD) in combination with optimized background therapy (OBT) (3 to 6 drugs based on treatment history and resistance testing). The 150 mg QD arm = placebo drug in the morning and active drug in the evening.
- Maraviroc BID: Maraviroc 150 mg PO twice a day (BID) in combination with OBT (3 to 6 drugs based on treatment history and resistance testing). The 150 mg BID arm = active drug in the morning and evening.
- Placebo: Placebo BID in combination with OBT (3 to 6 drugs based on treatment history and resistance testing). The placebo arm = placebo drug in the morning and evening.
Period: Assigned to Study Treatment
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Started | 63 | 63 | 64
Completed | 63 | 61 | 62
Not Completed | 0 | 2 | 2
Not completed — Randomized, but not treated | 0 | 2 | 2
Period: Received Study Treatment
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Started | 63 | 61 (Due to 1 placebo subject switched to maraviroc BID, BID = 62 subjects in Adverse event tables.) | 62 (Due to 1 placebo subject switched to maraviroc BID, Placebo = 61 subjects in Adverse event tables.)
Dual-tropic Subjects by Phenotype Assay | 57 (Dual-tropic: Virus capable of using both CCR5 and CXCR4 coreceptors for cell entry.) | 52 | 58
Completed | 15 | 25 | 18
Not Completed | 48 | 36 | 44
Not completed — Death | 2 | 1 | 2
Not completed — Adverse Event | 1 | 2 | 5
Not completed — Lack of Efficacy | 40 | 27 | 27
Not completed — Other | 2 | 2 | 6
Not completed — Subject defaulted | 3 | 4 | 4
Period: Continued on Open-Label Treatment
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Started | 15 | 25 | 0 (Placebo group not offered open-label maraviroc due to study not reaching primary endpoint at Week 24)
Completed | 7 | 10 | 0
Not Completed | 8 | 15 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Lack of Efficacy | 1 | 2 | 0
Not completed — Other reason includes protocol violation | 6 | 7 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo | Total
Number analyzed (Participants) | 63 | 61 | 62 | 186
Age, Customized [Number; unit: participants]
  <18 years | 2 | 2 | 0 | 4
  Between 18 and 24 years | 1 | 1 | 1 | 3
  Between 25 and 34 years | 2 | 3 | 2 | 7
  Between 35 and 44 years | 30 | 31 | 31 | 92
  Between 45 and 54 years | 25 | 21 | 20 | 66
  Between 55 and 64 years | 3 | 3 | 7 | 13
  ≥65 years | 0 | 0 | 1 | 1
Age Continuous [Mean (Full Range); unit: years] | 42.7 (8.4) [16 to 59] | 42.5 (8.0) [16 to 62] | 44.6 (8.3) [23 to 65] | 43.3 (8.2) [16 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 9 | 25
  Male | 53 | 55 | 53 | 161

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Human Immunodeficiency Virus (HIV-1) Viral Load (Ribonucleic Acid [RNA])
Description: Change from baseline in log 10-transformed plasma viral load (HIV-1 RNA) levels (log 10 copies per milliliter [log10 copies/mL]). Baseline value calculated as average of pre-dose measurements collected at screening, randomization, and baseline visits.
Time Frame: Baseline to Week 24 and Week 48
Population: Full Analysis Set (FAS)-as treated: all randomized subjects classified as dual-tropic by phenotype assay; received at least 1 dose of study treatment. Missing values: discontinuations (DC) imputed as baseline value (change from baseline=0); missing data imputed as Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Error); unit: log10 copies/mL
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Number analyzed (Participants) | 57 | 52 | 58
log10 copies/mL
  Week 24 | -0.890 (0.1706) | -1.194 (0.2060) | -0.953 (0.1795)
  Week 48 | -0.604 (0.1596) | -1.105 (0.2071) | 0.839 (0.1851)
Statistical Analysis 1: Comparison: Maraviroc QD vs Placebo; Maraviroc (MVC) QD versus placebo (PBO) treatment (TX) difference at Week 24. If upper bound of 97.5% confidence interval is <0, it is concluded that dose is superior to PBO. If upper bound is <0.25, it is concluded that MVC is non-inferior to PBO. Assumption: 79% of subjects are dual-tropic; total N=192 needed to be randomized to get N=150 dual-tropic. Standard deviation=0.8 with 2-sided p-value=0.025: 80% power for TX difference of 0.5 for change from baseline in log10-transformed viral load; Test type: Non-Inferiority or Equivalence — For hypothesis of superiority, if upper bound of 97.5% confidence interval (CI) of TX difference was <0 log10 copies/mL, it was concluded that MVC regimen was superior to PBO meaning that MVC added to Optimized Background Therapy (OBT) provides an additional reduction in plasma HIV-1 RNA compared to OBT alone. If superiority could not be concluded, then a hypothesis of noninferiority was tested. If upper bound of CI is <0.25 log10 copies/mL, noninferiority of MVC regimen to placebo was claimed; ANCOVA; TX difference adjusted for randomization strata. Bonferroni adjustment for multiple comparisons by use of 2-sided 97.5% CI to maintain alpha=0.05; Least squares mean = 0.055, 97.5% CI 2-sided [-0.528 to 0.638], Standard Error of Mean 0.2575 — Negative values for change from baseline=benefit of TX; negative values for MVC versus (vs) PBO=advantage of MVC
Statistical Analysis 2: Comparison: Maraviroc BID vs Placebo; MVC BID vs PBO treatment difference at Week 24; Test type: Superiority or Other; ANCOVA; [statistical method as in outcome 1, analysis 1]; Least squares mean = -0.232, 97.5% CI 2-sided [-0.829 to 0.364], Standard Error of Mean 0.2637 — Negative values for change from baseline=benefit of TX; negative values for MVC vs PBO=advantage of MVC
Statistical Analysis 3: Comparison: Maraviroc QD vs Placebo; MVC QD vs PBO treatment difference at Week 48; Test type: Superiority or Other; ANCOVA; [statistical method as in outcome 1, analysis 1]; Least squares mean = 0.229, 97.5% CI 2-sided [-0.351 to 0.810], Standard Error of Mean 0.2567 — Negative values for change from baseline=benefit of TX; negative values for MVC vs PBO=advantage of MVC
Statistical Analysis 4: Comparison: Maraviroc BID vs Placebo; MVC BID vs PBO treatment difference at Week 48; Test type: Superiority or Other; ANCOVA; [statistical method as in outcome 1, analysis 1]; Least squares mean = -0.261, 97.5% CI 2-sided [-0.856 to 0.333], Standard Error of Mean 0.2628 — Negative values for change from baseline=benefit of TX; negative values for MVC vs PBO=advantage of MVC

2. Secondary Outcome: Number of Subjects With HIV-1 RNA Levels < 400 Copies/mL
Time Frame: Week 24, Week 48
Population: FAS - as treated dual-tropic subjects. Missing values counted as failures/non-responders (counted as not achieving the stated criterion).
Measure: Number; unit: participants
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Number analyzed (Participants) | 57 | 52 | 58
participants
  Week 24 | 14 | 16 | 14
  Week 48 | 13 | 16 | 13
Statistical Analysis 1: Comparison: Maraviroc QD vs Placebo; MVC QD vs PBO treatment difference in proportions at Week 24; Test type: Superiority or Other; difference in proportions = 0.03, 95% CI 2-sided [-0.12 to 0.18] — The TX difference is weighted (by inverse of the variance) difference in proportions adjusted for randomization strata. Positive values for TX difference favor MVC. CI estimated using the normal approximation to the binomial distribution
Statistical Analysis 2: Comparison: Maraviroc BID vs Placebo; MVC BID vs PBO treatment difference in proportions at Week 24; Test type: Superiority or Other; difference in proportions = 0.07, 95% CI 2-sided [-0.08 to 0.23] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Maraviroc QD vs Placebo; MVC QD vs PBO treatment difference in proportions at Week 48; Test type: Superiority or Other; difference in proportions = 0.02, 95% CI 2-sided [-0.12 to 0.17] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Maraviroc BID vs Placebo; MVC BID vs PBO treatment difference in proportions at Week 48; Test type: Superiority or Other; difference in proportions = 0.09, 95% CI 2-sided [-0.07 to 0.25] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Number of Subjects With HIV-1 RNA Levels < 400 Copies/mL or at Least 0.5 Log 10-transformed Decrease From Baseline in HIV-1 RNA Levels
Description: Number of subjects with HIV-1 RNA levels < 400 copies/mL or at least 0.5 log 10-transformed decrease from baseline in HIV-1 RNA levels. Baseline value calculated as average of pre-dose measurements collected at screening, randomization, and baseline visits.
Time Frame: Baseline, Week 24, Week 48
Population: FAS-as treated dual-tropic subjects. Missing values counted as failures/non-responders (counted as not achieving the stated criterion).
Measure: Number; unit: participants
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Number analyzed (Participants) | 57 | 52 | 58
participants
  Week 24 | 24 | 25 | 23
  Week 48 | 14 | 22 | 18
Statistical Analysis 1: Comparison: Maraviroc QD vs Placebo; MVC QD vs PBO treatment difference in proportions at Week 24; Test type: Superiority or Other; difference in proportions = 0.03, 95% CI 2-sided [-0.15 to 0.20] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Maraviroc BID vs Placebo; MVC BID vs PBO treatment difference in proportions at Week 24; Test type: Superiority or Other; difference in proportions = 0.08, 95% CI 2-sided [-0.10 to 0.26] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Maraviroc QD vs Placebo; MVC QD vs PBO treatment difference in proportions at Week 48; Test type: Superiority or Other; difference in proportions = -0.06, 95% CI 2-sided [-0.22 to 0.10] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Maraviroc BID vs Placebo; MVC BID vs PBO treatment difference in proportions at Week 48; Test type: Superiority or Other; difference in proportions = 0.11, 95% CI 2-sided [-0.07 to 0.28] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Number of Subjects With HIV-1 RNA Levels < 400 Copies/mL or at Least 1.0 Log 10-transformed Decrease From Baseline in HIV-1 RNA Levels
Description: Number of subjects with HIV-1 RNA levels < 400 copies/mL or at least 1.0 log 10-transformed decrease from baseline in HIV-1 RNA levels. Baseline value calculated as average of pre-dose measurements collected at screening, randomization, and baseline visits.
Time Frame: Baseline, Week 24, Week 48
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Number analyzed (Participants) | 57 | 52 | 58
participants
  Week 24 | 18 | 23 | 21
  Week 48 | 13 | 20 | 15
Statistical Analysis 1: Comparison: Maraviroc QD vs Placebo; MVC QD vs PBO treatment difference in proportions at Week 24; Test type: Superiority or Other; difference in proportions = -0.05, 95% CI 2-sided [-0.21 to 0.12] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Maraviroc BID vs Placebo; MVC BID vs PBO treatment difference in proportions at Week 24; Test type: Superiority or Other; difference in proportions = 0.08, 95% CI 2-sided [-0.10 to 0.26] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Maraviroc QD vs Placebo; MVC QD vs PBO treatment difference in proportions at Week 48; Test type: Superiority or Other; difference in proportions = -0.02, 95% CI 2-sided [-0.18 to 0.13] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Maraviroc BID vs Placebo; MVC BID vs PBO treatment difference in proportions at Week 48; Test type: Superiority or Other; difference in proportions = 0.12, 95% CI 2-sided [-0.04 to 0.29] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Number of Subjects With HIV-1 RNA Levels < 50 Copies/mL
Time Frame: Baseline, Week 24, Week 48
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Number analyzed (Participants) | 57 | 52 | 58
participants
  Week 24 | 12 | 14 | 9
  Week 48 | 10 | 14 | 13
Statistical Analysis 1: Comparison: Maraviroc QD vs Placebo; MVC QD vs PBO treatment difference in proportions at Week 24; Test type: Superiority or Other; difference in proportions = 0.07, 95% CI 2-sided [-0.07 to 0.20] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Maraviroc BID vs Placebo; MVC BID vs PBO difference in proportions at Week 24; Test type: Superiority or Other; difference in proportions = 0.11, 95% CI 2-sided [-0.03 to 0.26] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Maraviroc QD vs Placebo; MVC QD vs PBO treatment difference in proportions at Week 48; Test type: Superiority or Other; difference in proportions = -0.04, 95% CI 2-sided [-0.18 to 0.10] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Maraviroc BID vs Placebo; MVC BID vs PBO treatment difference in proportions at Week 48; Test type: Superiority or Other; difference in proportions = 0.06, 95% CI 2-sided [-0.10 to 0.21] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Change From Baseline in CD4 Cell Count
Description: Change from baseline in CD4 cell count (measured as cells per microliter [cells/µL]). Baseline value calculated as the average of pre-dose measurements collected at screening, randomization, and baseline visits.
Time Frame: Baseline to Week 24 and Week 48
Population: FAS - as treated dual-tropic subjects. Placebo N: 4 subjects did not have on-treatment information. Missing data imputed using LOCF.
Measure: Mean (Standard Error); unit: cells/µL
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Number analyzed (Participants) | 57 | 52 | 54
cells/µL
  Week 24 | 59.237 (8.9661) | 62.651 (10.0234) | 36.367 (8.4477)
  Week 48 | 65.86 (10.822) | 78.87 (11.566) | 51.29 (12.523)
Statistical Analysis 1: Comparison: Maraviroc QD vs Placebo; MVC QD vs PBO treatment difference at Week 24; Test type: Superiority or Other; ANCOVA; TX difference adjusted for randomization strata; Least squares mean = 23.927, 95% CI 2-sided [-1.359 to 49.213], Standard Error of Mean 12.8025 — Negative values for change from baseline=benefit of TX; negative values for MVC vs PBO=advantage of MVC
Statistical Analysis 2: Comparison: Maraviroc BID vs Placebo; MVC BID vs PBO treatment difference at Week 24; Test type: Superiority or Other; ANCOVA; TX difference adjusted for randomization strata; Least squares mean = 26.679, 95% CI 2-sided [0.869 to 52.490], Standard Error of Mean 13.0678 — Negative values for change from baseline=benefit of TX; negative values for MVC vs PBO=advantage of MVC
Statistical Analysis 3: Comparison: Maraviroc QD vs Placebo; MVC QD vs PBO treatment difference at Week 48; Test type: Superiority or Other; ANCOVA; TX difference adjusted for randomization strata; Least squares mean = 14.61, 95% CI 2-sided [-17.80 to 47.03], Standard Error of Mean 16.412 — Negative values for change from baseline=benefit of TX; negative values for MVC vs PBO=advantage of MVC
Statistical Analysis 4: Comparison: Maraviroc BID vs Placebo; MVC BID vs PBO treatment difference at Week 48; Test type: Superiority or Other; ANCOVA; TX difference adjusted for randomization strata; Least squares mean = 27.71, 95% CI 2-sided [-5.38 to 60.80], Standard Error of Mean 16.754 — Negative values for change from baseline=benefit of TX; negative values for MVC vs PBO=advantage of MVC

7. Secondary Outcome: Change From Baseline in CD8 Cell Count
Description: Change from baseline in CD8 cell count (measured as cells/µL). Baseline value calculated as the average of pre-dose measurements collected at screening, randomization, and baseline visits.
Time Frame: Baseline to Week 24 and Week 48
Population: as for outcome 6
Measure: Mean (Standard Error); unit: cells/µL
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Number analyzed (Participants) | 57 | 52 | 54
cells/µL
  Week 24 | 391.061 (57.0135) | 322.683 (68.3315) | 154.293 (46.8100)
  Week 48 | 351.23 (54.653) | 342.87 (72.222) | 192.30 (62.578)
Statistical Analysis 1: Comparison: Maraviroc QD vs Placebo; MVC QD vs PBO treatment difference at Week 24; Test type: Superiority or Other; ANCOVA; TX difference adjusted for randomization strata; Least squares mean = 234.499, 95% CI 2-sided [74.913 to 394.084], Standard Error of Mean 80.7990 — Negative values for change from baseline=benefit of TX; negative values for MVC vs PBO=advantage of MVC
Statistical Analysis 2: Comparison: Maraviroc BID vs Placebo; MVC BID vs PBO treatment difference at Week 24; Test type: Superiority or Other; ANCOVA; TX difference adjusted for randomization strata; Least squares mean = 188.817, 95% CI 2-sided [23.999 to 353.635], Standard Error of Mean 83.4484 — Negative values for change from baseline=benefit of TX; negative values for MVC vs PBO=advantage of MVC
Statistical Analysis 3: Comparison: Maraviroc QD vs Placebo; MVC QD vs PBO treatment difference at Week 48; Test type: Superiority or Other; ANCOVA; TX difference adjusted for randomization strata; Least squares mean = 155.94, 95% CI 2-sided [-16.49 to 328.37], Standard Error of Mean 87.304 — Negative values for change from baseline=benefit of TX; negative values for MVC vs PBO=advantage of MVC
Statistical Analysis 4: Comparison: Maraviroc BID vs Placebo; MVC BID vs PBO treatment difference at Week 48; Test type: Superiority or Other; ANCOVA; TX difference adjusted for randomization strata; Least squares mean = 182.91, 95% CI 2-sided [4.81 to 361.02], Standard Error of Mean 90.174 — Negative values for change from baseline=benefit of TX; negative values for MVC vs PBO=advantage of MVC

8. Secondary Outcome: Time (50% Quartile Point Estimate) to Virologic Failure
Description: Time to virologic failure based on observed HIV-1 RNA levels and failure events (death; permanent discontinuation of test drug [perm DC]; lost to follow-up [LTFU]; new anti-retroviral drug added (except background drug change to drug of same class); or on open label for early non-response or rebound). Failure: at Time 0 if level not <400 copies/mL (2 consecutive visits) before event(s) or last available visit; at time of earliest event if level <400 copies/mL (on 2 consecutive visits); failure if level ≥400 copies/mL (2 consecutive visits) or 1 visit ≥400 copies/mL followed by perm DC or LTFU.
Time Frame: Day 1 through Week 24 and through Week 48
Population: FAS - as treated dual-tropic subjects; (n)=number of subjects with virologic failure at observation for maraviroc QD, maraviroc BID, and placebo, respectively; Week 48 result values (0.00)=virologic failure at Day 0.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Number analyzed (Participants) | 57 | 52 | 58
days
  Week 24 (n=35, 23, 29) | 88.00 [59.00 to NA] — Parameter was not calculable. | 189.00 [113.00 to 189.00] | 100.00 [60.00 to NA] — Parameter was not calculable.
  Week 48 (n=45, 37, 44) | 0.00 [NA to NA] — Parameters were not calculable. | 0.00 [0.00 to 142.00] | 0.00 [0.00 to 29.00]
Statistical Analysis 1: Comparison: Maraviroc QD vs Placebo; MVC QD vs PBO at Week 24. Kaplan-Meier survival estimates. TX difference evaluated by log-rank test; Test type: Superiority or Other; p = 0.7524, Log Rank
Statistical Analysis 2: Comparison: Maraviroc BID vs Placebo; MVC BID vs PBO at Week 24. Kaplan-Meier survival estimates. TX difference evaluated by log-rank test; Test type: Superiority or Other; p = 0.2540, Log Rank
Statistical Analysis 3: Comparison: Maraviroc QD vs Placebo; MVC QD vs PBO at Week 48. Kaplan-Meier survival estimates. TX difference evaluated by log-rank test; Test type: Superiority or Other; p = 0.8243, Log Rank
Statistical Analysis 4: Comparison: Maraviroc BID vs Placebo; MVC BID vs PBO at Week 48. Kaplan-Meier survival estimates. TX difference evaluated by log-rank test; Test type: Superiority or Other; p = 0.6657, Log Rank

9. Secondary Outcome: Change From Baseline in Time Averaged Difference (TAD) in log10 HIV-1 RNA
Description: Change from baseline of TAD in log10 HIV-1 RNA viral load calculated as [AUC of HIV-1 RNA viral load (log10 copies/mL) / time period] - Baseline HIV-1 RNA viral load (log10 copies/mL). Baseline value calculated as the average of pre-dose measurements collected at screening, randomization, and baseline visits.
Time Frame: Baseline to Week 24 and Week 48
Population: FAS - as treated dual-tropic subjects. Discontinuations prior to time point of analysis imputed as 0.
Measure: Mean (Standard Error); unit: log10 copies/mL
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Number analyzed (Participants) | 57 | 52 | 58
log10 copies/mL
  Week 24 | -0.850 (0.1510) | -1.151 (0.1895) | -0.926 (0.1679)
  Week 48 | -0.561 (0.1475) | -1.066 (0.1962) | -0.776 (0.1700)
Statistical Analysis 1: Comparison: Maraviroc QD vs Placebo; MVC QD vs PBO treatment difference at Week 24; Test type: Superiority or Other; ANCOVA; TX difference adjusted for randomization strata; Least squares mean = 0.069, 95% CI 2-sided [-0.396 to 0.535], Standard Error of Mean 0.2356
Statistical Analysis 2: Comparison: Maraviroc BID vs Placebo; MVC BID vs PBO treatment difference at Week 24; Test type: Superiority or Other; ANCOVA; TX difference adjusted for randomization strata; Least squares mean = -0.218, 95% CI 2-sided [-0.694 to 0.258], Standard Error of Mean 0.2413
Statistical Analysis 3: Comparison: Maraviroc QD vs Placebo; MVC QD vs PBO treatment difference at Week 48; Test type: Superiority or Other; ANCOVA; TX difference adjusted for randomization strata; Least squares mean = 0.209, 95% CI 2-sided [-0.262 to 0.681], Standard Error of Mean 0.2388
Statistical Analysis 4: Comparison: Maraviroc BID vs Placebo; MVC BID vs PBO treatment difference at Week 48; Test type: Superiority or Other; ANCOVA; TX difference adjusted for randomization strata; Least squares mean = -0.284, 95% CI 2-sided [-0.767 to 0.199], Standard Error of Mean 0.2445

10. Secondary Outcome: Number of Subjects Per Genotype and Phenotype at Baseline and at Time of Failure
Description: Number of subjects per genotype and phenotype (tests for presence of non CCR5-tropic HIV-1 and for resistance to reverse transcriptase, protease, and fusion inhibitors) at baseline and at time of failure through Week 48 visit. Sensitivity to drug categorized as 0-1, 2-4, >4; scores defined as 0=resistance, 1=sensitive or susceptible with higher number indicating greater sensitivity or susceptibility.
Time Frame: Baseline through Week 48
Population: FAS-as treated dual-tropic subjects. Genotype and phenotype at screening and at time of failure were not summarized as planned.
Measure: Number; unit: participants
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Number of Subjects Per Tropism Status at Screening and at the Time of Treatment Failure (Analysis at Week 24)
Description: Number of subjects per Tropism status (CCR5 [R5], CXCR4 [X4], Dual Mixed [DM], or Non-reportable/Non-phenotypable [NR/NP]) at Screening (Scr) and at time of treatment failure (Tx fail). Treatment failure defined as insufficient clinical response. HIV-1 RNA viral load <500 copies/ml categorized as below lower limit of quantification (BLQ). Tropism may have been assessed at either the Screening or Baseline visit. The assessment for time of treatment failure is defined as the last on-treatment assessment.
Time Frame: Screening through Week 24
Population: FAS-as treated; N=subjects with TX failure due to insufficient clinical response and who had a tropism assessment at Screening. Subjects with DC prior to timepoint not included; LOCF if no result (viral load too low for analysis).
Measure: Number; unit: participants
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Number analyzed (Participants) | 35 | 24 | 24
participants
  Scr: X4, Tx fail: X4 | 1 | 1 | 1
  Scr: X4, Tx fail: DM | 1 | 1 | 0
  Scr: DM, Tx fail: R5 | 1 | 0 | 4
  Scr: DM, Tx fail: X4 | 12 | 12 | 2
  Scr: DM, Tx fail: DM | 19 | 9 | 16
  Scr DM, Tx fail: NR/NP | 0 | 0 | 1
  Scr DM, Tx fail: BLQ | 1 | 0 | 0
  Scr NR/NP, Tx fail: NR/NP | 0 | 1 | 0

12. Secondary Outcome: Number of Subjects Per Tropism Status at Screening and Time of Treatment Failure (Analysis at Week 48)
Description: as for outcome 11
Time Frame: Screening through Week 48
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Number analyzed (Participants) | 40 | 27 | 27
participants
  Scr: X4, Tx fail: X4 | 1 | 1 | 1
  Scr: X4, Tx fail: DM | 1 | 1 | 0
  Scr: DM, Tx fail: R5 | 1 | 1 | 5
  Scr: DM, Tx fail: X4 | 12 | 12 | 2
  Scr: DM, Tx fail: DM | 24 | 10 | 18
  Scr: DM, Tx fail: NR/NP | 0 | 1 | 1
  Scr: DM, Tx fail: BLQ | 1 | 0 | 0
  Scr: NR/NP, Tx fail: NR/NP | 0 | 1 | 0

13. Secondary Outcome: Number of Subjects With Treatment Failure at Week 24 by Overall Susceptibility Score (OSS) at Screening
Description: Number of subjects for association between screening resistance and virologic response as determined by treatment failure and OSS at screening. OSS categorized as 0-1, 2-4, >4 (maximum value of 6) and calculated as the sum of the net assessment of in vitro phenotypic and genotypic susceptibility using a binary scoring system (0= reduced susceptibility, 1=susceptible) for each antiretroviral agent in OBT. Higher scores indicate greater susceptibility.
Time Frame: Screening, Week 24
Population: FAS - as treated dual-tropic subjects. Missing values imputed as LOCF.
Measure: Number; unit: participants
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Number analyzed (Participants) | 57 | 52 | 58
participants
  Scr score: 0-1 | 21 | 12 | 17
  Scr score: 2-4 | 35 | 35 | 40
  Scr score: missing | 1 | 1 | 1

14. Secondary Outcome: Number of Subjects With Treatment Failure at Week 48 by Overall Susceptibility Score (OSS) at Screening
Description: Number of subjects for association between screening resistance and virologic response as determined by treatment failure and OSS at screening. OSS categorized as 0, 1, 2, or ≥3 (maximum value of 6) and calculated as the sum of the net assessment of in vitro phenotypic and genotypic susceptibility using a binary scoring system (0= reduced susceptibility, 1=susceptible) for each antiretroviral agent in OBT. Higher scores indicate greater susceptibility.
Time Frame: Screening, Week48
Population: FAS - as treated dual-tropic subjects. Missing values imputed as LOCF.
Measure: Number; unit: particpants
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Number analyzed (Participants) | 57 | 52 | 58
particpants
  Scr score: 0 | 1 | 2 | 2
  Scr score: 1 | 19 | 11 | 15
  Scr score: 2 | 21 | 14 | 13
  Scr score: ≥3 | 15 | 24 | 27
  Scr score: missing | 1 | 1 | 1

15. Secondary Outcome: Number of Subjects With Acquired Immunodeficiency Syndrome (AIDS)-Defining Opportunistic Illnesses (Analysis at Week 24)
Description: Number of subjects with AIDS-defining opportunistic illnesses based on investigator classification guided by a predefined list of clinical Category C Adverse Events per Center for Disease Control (CDC) HIV Classification System. Includes events occurring up to 7 days after last dose of study drug.
Time Frame: Baseline through Week 24
Population: FAS - as randomized; N=number of subjects with Category C Adverse Events for maraviroc QD, maraviroc BID, and placebo, respectively. Week 48 results reflect subsequent updates to data originally reported at Week 24.
Measure: Number; unit: participants
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Number analyzed (Participants) | 63 | 61 | 62
participants
  Candidiasis | 0 | 0 | 1
  Cytomegalovirus chorioretinitis | 1 | 0 | 0
  Herpes simplex | 1 | 0 | 0
  Histoplasmosis | 1 | 0 | 0
  Mycobacterium avium complex infection | 1 | 0 | 0
  Oesophageal candidiasis | 0 | 2 | 0
  Pneumocystis jiroveci pneumonia | 3 | 1 | 0
  Pneumonia | 0 | 0 | 1
  Encephalitis | 0 | 0 | 1

16. Secondary Outcome: Number of Subjects With Acquired Immunodeficiency Syndrome (AIDS)-Defining Opportunistic Illnesses (Analysis at Week 48)
Description: Number of subjects with AIDS-defining opportunistic illnesses based on investigator classification guided by a predefined list of clinical Category C Adverse Events per CDC HIV Classification System. Includes events occurring up to 7 days after last dose of study drug.
Time Frame: Baseline through Week 48
Population: as for outcome 15
Measure: Number; unit: participants
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Number analyzed (Participants) | 63 | 61 | 62
participants
  Candidiasis | 0 | 1 | 1
  Cytomegalovirus chorioretinitis | 1 | 0 | 0
  Histoplasmosis | 1 | 0 | 0
  Oesophageal candidiasis | 0 | 2 | 0
  Pneumococcal Sepsis | 0 | 1 | 0
  Pneumocystis jiroveci pneumonia | 3 | 0 | 0
  Pneumonia | 0 | 1 | 0
  Encephalitis | 0 | 0 | 1

ADVERSE EVENTS:
Arm/Group | Maraviroc QD | Maraviroc BID | Placebo
Serious Adverse Events (participants affected / at risk) | 13/63 | 14/62 | 13/61
Other Adverse Events (participants affected / at risk) | 46/63 | 51/62 | 42/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Maraviroc QD (N=63) | Maraviroc BID (N=62) | Placebo (N=61)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 1
Condition aggravated (General disorders) | 0 | 0 | 1
Disease progression (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 3 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 1
Abscess (Infections and infestations) | 0 | 0 | 1
Bronchitis bacterial (Infections and infestations) | 0 | 0 | 1
Candidiasis (Infections and infestations) | 0 | 0 | 1
Clostridial infection (Infections and infestations) | 0 | 2 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Histoplasmosis (Infections and infestations) | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 1
Meningitis aseptic (Infections and infestations) | 1 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 2 | 0
Pneumococcal sepsis (Infections and infestations) | 0 | 1 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 3 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 2 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Staphylococcal abscess (Infections and infestations) | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Central nervous system lesion (Nervous system disorders) | 0 | 0 | 1
Encephalitis (Nervous system disorders) | 0 | 0 | 1
Movement disorder (Nervous system disorders) | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 2
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Maraviroc QD (N=63) | Maraviroc BID (N=62) | Placebo (N=61)
Anaemia (Blood and lymphatic system disorders) | 4 | 0 | 1
Constipation (Gastrointestinal disorders) | 6 | 5 | 1
Diarrhoea (Gastrointestinal disorders) | 18 | 12 | 13
Nausea (Gastrointestinal disorders) | 9 | 8 | 12
Vomiting (Gastrointestinal disorders) | 8 | 3 | 8
Asthenia (General disorders) | 0 | 2 | 7
Fatigue (General disorders) | 8 | 10 | 11
Injection site reaction (General disorders) | 7 | 13 | 9
Pyrexia (General disorders) | 5 | 6 | 4
Bronchitis (Infections and infestations) | 4 | 6 | 2
Herpes simplex (Infections and infestations) | 4 | 4 | 2
Influenza (Infections and infestations) | 1 | 4 | 1
Nasopharyngitis (Infections and infestations) | 5 | 3 | 3
Oral candidiasis (Infections and infestations) | 1 | 5 | 0
Pharyngitis (Infections and infestations) | 1 | 5 | 0
Sinusitis (Infections and infestations) | 3 | 6 | 4
Upper respiratory tract infection (Infections and infestations) | 5 | 10 | 5
Weight increased (Investigations) | 4 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 8 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 6 | 2
Dizziness (Nervous system disorders) | 6 | 6 | 3
Headache (Nervous system disorders) | 13 | 11 | 5
Insomnia (Psychiatric disorders) | 5 | 5 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 4 | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3 | 5
Rash (Skin and subcutaneous tissue disorders) | 7 | 6 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.